CLINICAL TRIAL: NCT04896463
Title: Comparative Study of FAST (Focussed Assessment With Sonography in Trauma) Versus Multidetector Computed Tomography (CT) Scan of the Abdomen in Patients With Abdominal Trauma
Brief Title: Comparative Study of FAST Versus Multidetector CT Scan of the Abdomen in Patients With Abdominal Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Salah El-Dein Quashty Aly, Emergency medicine resident physician, Assiut University
Other Study IDs: FAST
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: FAST (Focussed Assessment With Sonography in Trauma)
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Abdominal ultrasound (US) — abdominal examination with US device
  Other Names: multidetector computed tomography (CT) scan of the abdomen

SUMMARY:
The aim of the study is to evaluate the diagnostic accuracy of FAST (as regards sensitivity and specificity) as an initial assessment for patients with abdominal trauma compared to that of the gold standard multidetector CT scan of the abdomen.

DETAILED DESCRIPTION:
Trauma is a major health problem in every country, regardless of the level of socioeconomic development, associated with high morbidity and mortality as it is still the most frequent cause of death in the first four decades of life.According to the World Health Organization, more than nine people die per minute victimized by trauma, It is costy on the health services more than other diseases with a rate upto 12%.

In Egypt the mortality from road traffic crashes is about 12000 victims per year, with fatality rate of about 42 deaths per 100 000 population. Majority (48%) of them are passengers of motor vehicles. Car accidents in Egypt rose by 17.8% in 2019 with 9,992 compared to 8,480 in 2018 that is announced by The Central Agency For Public Mobilization and Statistics (CAPMAS).

The abdomen is the third most common injured region with surgery required in about 25% of civilian cases.

Abdominal trauma is traditionally classified as either blunt or penetrating (stab or gunshot wounds) which can usually be diagnosed easily and reliably, whereas blunt abdominal trauma is often missed because clinical signs are less obvious.Blunt abdominal injuries predominate in rural areas, while penetrating ones are more frequent in urban settings.

In order to minimize mortality in cases of abdominal trauma, risk factors for mortality needed to be systematically identified and studied. In recent years studies have identified a number of such risk factors, including sex, the length of the interval between abdominal injury and surgery, shock at the time of admission, and cranial injuries.

So appropriate care of the trauma patient entails a multidisciplinary effort that requires speed, efficiency,and proper coordination of the initial care team to make fast rational decisions.In such patient focussed abdominal ultrasonograpghy (FAST) often is the initial imaging examination.

FAST is readily available , low cost, repeatable noninvasive bedside method ,requires minimal preparation time ,and may be performed with mobile equipment that allows greater flexibility in patient positioning than is possible with other imaging modalities .It is also effective in depicting abnormally large intraperitoneal collections of free fluid, which are indirect evidence of a solid organ injury that requires emergency laparotomy.

However, not all clinically important abdominal injuries have associated hemoperitoneum such as those to the bowel , diaphragm, and mesentery. So an initial survey with FAST is often followed by a more thorough examination with multidetector computed tomography (CT) which became the imaging modality of choice in the late 1990s.It is a useful sen e method to detect intraperitoneal free air and intraperitoneal fluid,delineate the extent of solid organ injury,detect retroperitoneal injuries, and help in the decision of conservative nonsurgical therapy.But the adverse effects of it are that it is time consuming procedure and not advisable in hemodynamically unstable patients, moreover it is expensive and carries high risk of radiation exposure when repeated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged ≥18 years).
2. Patients exposed to different mechanisms of abdominal trauma whether penetrating such as : stab or gunshot wounds . Or a blunt mechanism of trauma such as:motor vehicle collisions ,falls from height ,assaults ,falling down , falling a heavy object on torso , and sports accidents .

Exclusion Criteria:

1. Pregnant females.
2. Any patient who undergoes urgent surgical intervention as a primary survey.
3. Patient refusal to participate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: : The study will be conducted on patients admitted with abdominal trauma in Assuit or Alexandria Main University Hospitals after obtaining their or their next of kin consent to participate in the study without affecting their course of treatment according to permission obtained from ethical committee of faculty of medicine in Assiut and Alexandria universities.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
The presence (positive FAST) or absence (negative FAST) of intraperitoneal free fluid collection in the four standard views to ascertain accuracy of FAST as regards sensitivity and specificity. | baseline
  : FAST examination is performed using a mobile US machine with a curvilinear 3.5 to 5 -MHz probe while the patient in a recumbent position and the examiner stands to the right of the patient to obtain the following four standard views:
  * Transverse view of the subxiphoid region to assess the pericardial space and injuries to the left lobe of the liver.
  * Longituidinal view of the right upper quadrant (RUQ) to show the right lobe of the liver, the right kidney, the space between the two(the Morison pouch), and the right paracolic gutter.
  * Longituidinal view of the left upper quadrant (LUQ) to show the left kidney, the spleen, the space between them, and the left para colic gutter.
  * Transverse and longituidinal views of the suprapubic region to depict the urinary bladder and rectouterina or retrovesical pouch.

IPD SHARING:
Plan to Share IPD: Undecided